CLINICAL TRIAL: NCT01179113
Title: Esmolol Infusion for Maintaining Hemodynamic Stability During Single or Double Level Lumbar Laminectomy: Effect on Quality of Recovery.
Brief Title: Esmolol Infusion During Laminectomy: Effect on Quality of Recovery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The preliminary result didn't show any benefit.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Roya Yumul, M.D.,PhD., Residency program director, Department of anesthesiology, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Pro00019850
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Results first posted 2016-08-30 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-09

CONDITIONS: Laminectomy
Keywords: Laminectomy; Esmolol Infusion; Quality of recovery; beta-blockers; Pain management; Postoperative pain; Opioid requirements; Intraoperative esmolol infusion; Return to normal activities of daily living
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — esmolol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo: Will receive a normal saline bolus during induction, and an infusion of normal saline intraoperatively
  Interventions: Drug: Saline
- Esmolol (Active Comparator): Will receive Esmolol Loading: 0.5 mg/kg bolus during induction Infusion: 15 mcg /kg/min, infusion intraoperatively
  Interventions: Drug: Esmolol

INTERVENTIONS:
Drug: Esmolol — Esmolol group: Will receive 0.5 mg/kg IV bolus of esmolol during induction, and an infusion of esmolol at 0.3 mg/kg/hr intraoperatively.
  Other Names: Brevibloc
  Arms: Esmolol
Drug: Saline — Loading: an equivalent volume for the Esmolol group Infusion: an equivalent volume for the Esmolol group
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of esmolol, a drug which is commonly administered during surgery to help control blood pressure and heart rate, on postoperative pain levels and requirements for pain medication.

DETAILED DESCRIPTION:
A common practice used to control autonomic responses during surgery is to administer beta-blockers intraoperatively. This practice has been shown to effectively blunt autonomic responses to intraoperative events. Several studies have shown that administration of beta-blockers can decrease intraoperative anesthetic requirements. Additionally, it has been demonstrated in several studies that intraoperative beta-blocker administration may actually decrease postoperative pain scores and opioid requirements, although these results are not entirely consistent. The mechanism by which the decrease in postoperative pain and narcotic requirements occurs is unclear. It has been postulated that esmolol may itself possess some analgesic-like properties, as was suggested by studies performed in rodent models. It has also been postulated that perioperative beta-blockade may attenuate the neuroendocrine stress response to surgery, thereby decreasing inflammatory responses in tissues; however, this theory was not supported by a study in which stress hormone levels were measured in patients who received beta-blockers and compared to a control group. Several studies which investigated the effects of beta-blockade on postoperative pain and opioid requirements compared the beta-blocker treatment group to an opioid treatment group, and did not include a true control group in which no treatment was given. Therefore, it is unclear whether the decrease in postoperative pain and opioid requirements in these studies was due to a true effect of the beta-blockers or whether it was due to an effect of the opioids.

Therefore, the investigators propose a randomized, double-blinded, placebo-controlled study in which the investigators will compare an esmolol infusion treatment group to a normal saline infusion control group with regards to the effects on postoperative pain and opioid requirements. By setting up the study in this manner, the investigators will be able to clearly evaluate the effects of beta-blockers on postoperative pain scores and opioid requirements. The investigators chose to use esmolol both because it has a short half-life, so it is easy to titrate and administer as an infusion, and also because it is selective for beta-1 receptors, so deleterious effects of intraoperative hypotension should be minimized. The investigators chose to perform the study on patients who are undergoing single-level or double-level laminectomies because prior studies have investigated the effects of intraoperative beta-blockers on patients who are not chronic pain patients, and the investigators would like to research whether the results which have been suggested by prior studies are also applicable to patients who may have chronic pain, as this is the patients population that is most likely to experience high pain levels following surgery, and may benefit the most from reduction of postoperative pain levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo single-level or double-level laminectomy under general anesthesia
* Willingness and ability to sign an informed consent document
* No allergies to any of the anesthetic or analgesic medications being used for the study, as outlined in the study protocol
* Between 18-80 years of age
* American Society of Anesthesiologists (ASA) class I-III adults of either sex

Exclusion Criteria:

* Patients who are ASA class IV or higher
* Patients with known allergy, hypersensitivity, or contraindication to the use of any of the medications being used for the study, as outlined in the study protocol
* Patients who are heavy chronic opioid users, defined for the purposes of this study as any patient who is taking the equivalent of 10mg of oral morphine per day or greater
* Pregnant or lactating women
* Patients with a history of drug or alcohol abuse within the past 3 months
* Patients with any other medical conditions or who are using any medications which may interfere with the conduct of the study (including patients taking clonidine, patients with EKG conduction defects and who are taking calcium channel blockers, patients with clinically significant congestive heart failure (CHF) or bronchospasm, or patients with second- or third-degree heart block, symptomatic sinus bradyarrhythmia, or nonsinus rhythm on preoperative EKG.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roya Yumul, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center; Roya Yumul, MD., PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to the day of surgery, potential study patients scheduled to undergo spine surgical procedures received a packet of materials from their surgeon. The packet contained an initial patient contact letter, a privacy information sheet, and the institution review board (IRB)-approved informed consent form.
Groups:
- Placebo: A normal saline bolus during induction, and an infusion of normal saline intraoperatively.
- Esmolol: Loading: 0.5 mg/kg bolus during induction Infusion: 15 mcg /kg/min, infusion intraoperatively
Period: Overall Study
Arm/Group | Placebo | Esmolol
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Esmolol | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (11) | 54 (16) | 57 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26 (5) | 26 (4) | 26 (5)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Using Verbal Rating Scale (VRS)
Description: Verbal Rating Scale goes from 0 to 10, where:
  0 indicates= No pain" and 10 indicates= The worst possible pain
  The information was be recorded by study staff and data obtained from patient and patient charts from post-anesthesia care unit (PACU) stay
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Esmolol
Number analyzed (Participants) | 17 | 16
Scores on a scale | 4 (4) | 5 (3)

2. Secondary Outcome: Opioid Consumption in PACU Obtained From the Recorded Data
Description: Postoperative use of opioid (Hydromorphone) consumption inside hospital at PACU (recorded by study staff and data obtained from patient charts).
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Placebo | Esmolol
Number analyzed (Participants) | 17 | 16
mg | 1.5 (0.6) | 2 (2.6)

3. Secondary Outcome: Postoperative Nausea and Vomiting
Description: Number of participants that experienced Postoperative nausea and vomiting using at PACU
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Placebo | Esmolol
Number analyzed (Participants) | 17 | 16
participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Placebo | Esmolol
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No